CLINICAL TRIAL: NCT05068674
Title: A Phase I, Randomized Pilot Study of Human Embryonic Stem Cell-Derived Cardiomyocytes (hESC-CMs) in PaTients With ChrOnic Ischemic Left VentRicular Dysfunction Secondary to Myocardial Infarction (HECTOR)
Brief Title: Human Embryonic Stem Cell-Derived Cardiomyocyte Therapy for Chronic Ischemic Left Ventricular Dysfunction
Acronym: HECTOR
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Joseph C. Wu (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor-Investigator, Joseph C. Wu, Professor of Medicine and Radiology., Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 60978
Record Dates: First submitted 2021-09-24; First posted 2021-10-06 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Chronic Ischemic Left Ventricular Dysfunction
MeSH Terms: interventions — Cell Count

STUDY DESIGN:
Intervention Model Description: Phase I will be a standard 3+3 dose-escalation study to evaluate 3 doses of allogeneic hESC-CMs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Active Comparator): Low dose (50M cells)
  Interventions: Drug: Human Embryonic Stem Cell-Derived Cardiomyocyte 50M cells
- Cohort 2 (Active Comparator): Medium dose (150M cells)
  Interventions: Drug: Human Embryonic Stem Cell-Derived Cardiomyocyte 150 cells
- Cohort 3 (Active Comparator): High dose (300M cells)
  Interventions: Drug: Human Embryonic Stem Cell-Derived Cardiomyocyte 300M cells

INTERVENTIONS:
Drug: Human Embryonic Stem Cell-Derived Cardiomyocyte 50M cells — 50 million (M) cells delivered in a dose of 5M cells per injection over 10 injections.
  Other Names: Human ESC-CMs
  Arms: Cohort 1
Drug: Human Embryonic Stem Cell-Derived Cardiomyocyte 150 cells — 150M cells delivered in a dose of 15M cells per injection over 10 injections
  Other Names: Human ESC-CMs
  Arms: Cohort 2
Drug: Human Embryonic Stem Cell-Derived Cardiomyocyte 300M cells — 300M cells delivered in a dose of 30M per injection over 10 injections
  Other Names: Human ESC-CMs
  Arms: Cohort 3

SUMMARY:
This clinical study will utilize a new cell therapy approach (Human embryonic stem cells derived cardiomyocytes or hESC-CMs) to improve survival and cardiac function in patients with chronic left ventricular dysfunction secondary to MI (Myocardial Infarction).

DETAILED DESCRIPTION:
The phase I dose-escalation pilot study is intended as an initial safety assessment to establish the MTD prior to the phase II randomized, double-blinded, placebo-controlled study. An estimated eighteen (18) patients in phase I who are scheduled to undergo cardiac catheterization and have met all inclusion/exclusion criteria will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥ 21 and < 80 years of age.
* Provide written informed consent.
* Have a diagnosis of chronic ischemic left ventricular dysfunction secondary to MI as defined by previous myocardial infarction documented by an imaging study demonstrating coronary artery disease with corresponding areas of akinesis, dyskinesis, or severe hypokinesis.
* Be a candidate for cardiac catheterization within 5 to 10 weeks of screening.
* Have been treated with appropriate maximal medical therapy for heart failure or postinfarction left ventricular dysfunction. For beta-blockade, the patient must have been on a stable dose of a clinically appropriate beta-blocker for 3 months. For angiotensinconverting enzyme (ACE) inhibitors or angiotensin receptor blockers (ARBs) or angiotensin receptor neprilysin inhibitors (ARNIs) or have appropriate medical indication precluding use of one or both of these agents, the patient must have been on a stable dose of a clinically appropriate agent for 1 month or within no more than doubling the dose of any of ARB, ACE inhibitors, and ARNIs over the last 3 months.
* Left ventricular ejection fraction below 40%.
* Class II/III NYHA symptoms of heart failure within the 6 months prior to baseline testing.
* Hospitalization in the past 6 months or NT pro-BNP > 1200 pg/mL, or >1600 pg/mL if atrial fibrillation was present.
* Automated implantable cardioverter-defibrillator (AICD) in place.

Exclusion Criteria:

* Have a baseline glomerular filtration rate < 35 ml/min/1.73 m2
* Have a known, serious radiographic contrast allergy.
* Have a prosthetic aortic valve or heart constrictive device.
* Have a documented presence of aortic stenosis (aortic stenosis graded as 1.5 cm2 or less).
* Have a documented presence of moderate to severe aortic insufficiency (echocardiographic assessment of aortic insufficiency graded as ≥+2).
* Have evidence of a life-threatening arrhythmia in the absence of a defibrillator (nonsustained ventricular tachycardia ≥ 20 consecutive beats or complete second- or third-degree heart block in the absence of a functioning pacemaker) or QTc interval > 550 ms on screening ECG.
* AICD firing in the past 60 days prior to enrollment.
* Be eligible for or require coronary artery revascularization.
* Have a hematologic abnormality as evidenced by hematocrit < 25%, white blood cell < 2,500/µl, or platelet values < 100,000/µl without another explanation.
* Have liver dysfunction, as evidenced by enzymes (AST and ALT) greater than three times the ULN.
* Have a coagulopathy (INR > 1.3) not due to a reversible cause (i.e., Coumadin). Patients on Coumadin will be withdrawn 5 days before the procedure and confirmed to have an INR < 1.3. Patients who cannot be withdrawn from Coumadin will be excluded from enrollment.
* Have known allergies to penicillin or streptomycin.
* Be an organ transplant recipient.
* Have a history of organ or cell transplant rejection.
* Have a clinical history of malignancy within 5 years (i.e., patients with prior malignancy must be disease-free for 5 years), except curatively-treated basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma.
* Have a non-cardiac condition that limits lifespan to < 1 year.
* Be on chronic therapy with immunosuppressant medication, such as corticosteroids or TNFα antagonists.
* Be serum-positive for HIV, hepatitis BsAg, or viremic hepatitis C.
* Be currently participating (or participated within the previous 30 days) in an investigational therapeutic or device trial.
* Be a female patient who is pregnant, nursing, or have child-bearing potential but is not using effective birth control.
* Tested positive for SARS-CoV-2 within the last 30 days

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) among 3 dose levels of allogeneic human embryonic stem cell-derived cardiomyocytes (hESC-CMs) | 3 Years
  The primary endpoints are safety and feasibility. The feasibility of preparing and delivering the study product, as well as collecting cardiac MRI variables in subjects will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Hospital and Clinics, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No